CLINICAL TRIAL: NCT05348928
Title: A Pilot Study of the Feasibility and Accuracy of the TrueVie Continuous Glucose Monitoring System - A Non-Significant Risk Study
Brief Title: A Pilot Study of the Feasibility and Accuracy of the TrueVie CGM System - A Non-Significant Risk Study
Status: Completed | Type: Observational
Sponsor: Sinocare Meditech Inc. (Industry)
Collaborators: Integrated Medical Development (Industry)
Responsible Party: Sponsor
Organization: Sinocare (Industry)
Other Study IDs: NPI031-CEP-001F
Record Dates: First submitted 2022-04-14; First posted 2022-04-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-05

CONDITIONS: Continuous Glucose Monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- With oral ascorbic acid: 1 g ascorbic acid orally
  Interventions: Device: Continuous glucose monitoring device; Other: Laboratory plasma glucose concentration determination
- Without oral ascorbic acid: No oral ascorbic acid is taken
  Interventions: Device: Continuous glucose monitoring device; Other: Laboratory plasma glucose concentration determination

INTERVENTIONS:
Device: Continuous glucose monitoring device — Continuous glucose monitoring device
Other: Laboratory plasma glucose concentration determination — Laboratory plasma glucose concentration determination

SUMMARY:
The purpose of the investigation is to obtain sufficient preliminary information about the performance of the TrueVie Continuous Glucose Monitoring (CGM) device to identify any need for any design modifications.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will be screened for participation. Qualifying participants will insert CGM sensors and come to 3 clinic visits at the beginning, middle and end of the 15 days intended sensor life. At the clinic visits participants are served two meals and perform a brief period of exercise of moderate intensity while blood samples are drawn according to a planned schedule timed to coincide with the TrueVie measurements.

ELIGIBILITY:
Inclusion Criteria:

1 Type 1 diabetes mellitus 2. Must be and have been in stable treatment regimen for at least 3 months with a multiple daily insulin dosing regimens or Continuous Subcutaneous Insulin Infusion (CSII), irrespective of delivery device(s).

3. Must have normal exercise tolerance.

Exclusion Criteria:

1. Skin adhesive tolerance issues in the area of sensor placement
2. HbA1c > 9%.
3. Insulin meal dosing based on fixed dose regimens.
4. Absence of established corrective factor for high glucose.
5. Hematocrit below 10% under the lower limit of the normal range.
6. Body mass index < 20 kg/m2.
7. Inadequate intravenous access on arms.
8. Absence of moderate exercise tolerance per history
9. Pregnancy, planned pregnancy within the study period, or unwillingness to use reliable contraception during the study period.
10. Planned MRI, CT scan or diathermic procedure for the duration of the study.
11. Any medical history of malignant melanoma or breast cancer.
12. Medical history of any other cancers within the last five years except adequately treated basal cell or squamous carcinoma of the skin, or cervical carcinoma in-situ.
13. History of alcohol or drug abuse within the last year.
14. Any condition that in the opinion of the investigator may interfere successful completion of study procedures.
15. Participation in other clinical trials involving receipt of investigational drug that cannot be disclosed within the last 30 days.
16. Inability or unwillingness to conform to the required protocol procedures including giving informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 15 days
  safety is assessed by adverse events
Incidence of Treatment-Emergent Adverse Device Events | 15 days
  safety is assessed by adverse device effects
Insertion Site Intensity of any Erythema on a Likert scale | 15 days
  tolerability by intensity of erythema at the insertion site
Insertion Site Erythema Size estimated from Lengths of Major and Minor Axis | 15 days
  tolerability by size of erythema at the insertion site
Edema by Maximal Height from Surrounding Skin Surface | 15 days
  tolerability by edema at insertion site

SECONDARY OUTCOMES:
Sensor Accuracy by Mean Absolute Glucose Concentration Difference from Reference | 15 days
  Sensor accuracy will be determined against plasma glucose concentrations determined by laboratory quality instrumentation

CONTACTS AND LOCATIONS:
Overall Officials: Poul Strange, MD, PhD, Study Director — Integrated Medical Development
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No